CLINICAL TRIAL: NCT07242079
Title: Effect of Pulmonary Rehabilitation and Physical Activity in Patients With Alpha-1 Antitrypsin Deficiency
Brief Title: Effect Of Pulmonary Rehabilitation in Patients With Alpha-1 Antitrypsin Deficiency
Acronym: RRALFA1
Status: Completed | Type: Observational
Sponsor: University of Parma (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 31276
Record Dates: First submitted 2025-06-27; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-07

CONDITIONS: Alpha-1 Antitrypsin Deficiency (AATD)
Keywords: Alpha-1 antitrypsin deficiency; Pulmonary rehabilitation; Active Cycle of Breathing Technique
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with alpha-1 antitrypsin deficiency (AATD): Adults with a confirmed diagnosis of alpha-1 antitrypsin deficiency (AATD) with asthma and/or COPD.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — the Active Cycle of Breathing Technique (ACBT) is a simple, standardized, and home-based technique that patients can perform with or without digital tools. ACBT has already been shown to improve forced vital capacity, peak expiratory flow, arterial oxygenation and exercise capacity.

SUMMARY:
This single-center, longitudinal, observational, prospective study aims to assess the applicability, adherence, and clinical impact of the Active Cycle of Breathing Technique (ACBT) with augmented reality support in patients with alpha-1 antitrypsin deficiency (AATD).

A total of 50 adult AATD patients will be recruit from the Lung Function Unit of the University Hospital of Parma, meeting specific inclusion criteria. Participants will perform ACBT twice daily and walk at least 5000 steps per day. Clinical and functional outcomes including dyspnea perception, lung function, and quality of life, will be assessed before and after a six-week ACBT program.

The study explores whether augmented reality enhance adherence and efficacy compared to conventional pulmonary rehabilitation (PR) methods. The expected outcome is improved adherence to PR.

DETAILED DESCRIPTION:
Alpha-1 antitrypsin deficiency (AATD) is a genetic disorder caused by mutations in the SERPINA1 gene, located on chromosome 14. The condition is characterized by low circulating levels of alpha-1 antitrypsin (AAT), a glycoprotein primarily produced by hepatocytes, which plays a crucial role in inhibiting neutrophil elastase (NE). Without adequate AAT, unregulated NE activity damages the lung parenchyma, leading to progressive emphysema. AATD presents with variable phenotypic expression, ranging from asymptomatic individuals to those with severe pulmonary and hepatic complications.

Treatment includes intravenous AAT replacement therapy, vaccination and guideline-recommended pulmonary rehabilitation (PR) based on the patient's clinical condition.

PR consists of a structured program combining breathing exercises, physical training, education, and psychological support to optimize respiratory function and improve patients' quality of life. One of the most effective techniques within PR is the Active Cycle of Breathing Technique (ACBT), which enhances airway clearance and lung function. ACBT is a simple, standardized, and home-based technique that patients can perform with or without digital tools. ACBT has already been shown to improve forced vital capacity, peak expiratory flow, arterial oxygenation and exercise capacity.

A tendency towards poor adherence to PR has been reported in the literature. To facilitate the performance of PR procedures, technological evolution in recent decades has brought new complementary techniques such as active video games, virtual reality and augmented reality.

ThIs study aims to assess satisfaction, adherence, and usability of pulmonary rehabilitation techniques in AATD patients, both with and without technological support, through relevant questionnaires (VAS, RAI, USE, TAM). Additionally, it aims to describe changes in the perception of dyspnea (mMRC), quality of life (EuroQol 5), impact of the pathology on daily life, and some functional parameters (FEV1, FVC, R5-R20, LCI, metres walked assessed by the six-minute walking test) at baseline and at the end of the rehabilitation program.

Data will be collected in a dedicated electronic Clinical Records Form (CRF). The database will be saved on a password-protected company Personal Computer (PC) which will be updated at each visit and used exclusively for scientific research purposes. At the time of enrollment, each patient will receive an alphanumeric code so that any information collected during the study, and in particular sensitive data, is treated in an anonymous manner. Data reporting patients' identifications will only be used to file patients and collect informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥18 years;
* Signed informed consent;
* All AATD patients, regardless of nephelometric alpha-1 antitrypsin dose and clinical phenotype, who require PR according to guidelines

Exclusion Criteria:

* Subjects unable to perform the lung function tests and rehabilitation program required by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of 50 adult patients, referred at outpatient clinic of the Respiratory Disease Unit of the University Hospital of Parma (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with PR techniques using Technology Acceptance Model (TAM) questionnaire. | six weeks
  Satisfaction will be assessed using the Technology Acceptance Model (TAM) questionnaire, with scores ranging from 1 to 7, where lower scores indicate more satisfaction.
Patient adherence to the PR techniques using the Rehabilitation Adherence Index (RAI) questionnaire. | six weeks
  Adherence will be assessed using the Rehabilitation Adherence Index (RAI) questionnaire, with scores ranging from 1 to 7, where higher scores indicate better adherence.
Usability of pulmonary rehabilitation techniques using the Usefulness, Satisfaction and Ease of Use (USE) questionnaire | six weeks
  Usability will be measured using the Usefulness, Satisfaction and Ease of Use (USE) questionnaire, with scores ranging from 1 to 7, where higher scores indicate better usability.

SECONDARY OUTCOMES:
To describe the change in perception of dyspnea at baseline and at the end of the PR using Modified Medical Research Council (mMRC) questionnaire. | six weeks
  The Modified Medical Research Council (mMRC) questionnaire assesses the perception of dyspnea with scores ranging from 0 to 4, with higher scores indicating greater severity.
To describe the change in quality of life at baseline and at the end of the PR using EuroQol-5D (EQ-5D) questionnaire. | six weeks
  The EQ-5D questionnaire assesses health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity: no problems, slight problems, moderate problems, severe problems, and unable to perform/extreme problems. Additionally, the EQ-5D includes a visual analogue scale (VAS) where respondents rate their overall health on a scale from 0 to 100, with 0 being the worst imaginable health and 100 being the best.
To assess the impact of Chronic Obstructive Pulmonary Disease (COPD) on AATD- related COPD patients using COPD Assessment Test (CAT) | six weeks
  The COPD Assessment Test (CAT) is assess the impact of Chronic Obstructive Pulmonary Disease (COPD) on a person's daily life. It ranges from 0 to 5, where higher scores indicate a greater impact of COPD on daily life
To assess the impact of asthma on AATD patients with asthma using the Asthma Control Test (ACT) | six weeks
  The Asthma Control Test (ACT) is a questionnaire used to assess asthma control, with scores ranging from 5 to 25. Higher scores indicate better asthma control, meaning the asthma is well-managed and less likely to interfere with daily activities.
To describe the change in functional respiratory parameters at baseline and at the end of the PR program using spirometry. | six weeks
  Spirometry will be performed according to ATS/ERS standards to obtain Forced Expiratory Volume in 1 second (FEV₁, % predicted), Forced Vital Capacity (FVC, % predicted), and FEV₁/FVC, %.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma, Parma, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected in a dedicated electronic Clinical Records Form (CRF). The database will be saved on a password- protected company personal computer which will be updated at each visit and used exclusively for scientific research purposes. At the time of enrolment, each patient will receive an alphanumeric code so that any information collected during the study, and in particular sensitive data, will be treated in an anonymous manner. Data reporting patients' identifications will only be used to file patients and collect informed consent.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available during the course of the study. The Investigator will keep paper and electronic copies of all documentation at the Center for a period of at least 7 years after the completion of the study and then he will arrange for its destruction.
Access Criteria: Only the personal delegated to collaborate with this study will be able to access to the database using a password to login.

REFERENCES:
- [Result] Conrad A, Janciauskiene S, Kohnlein T, Fuge J, Ivanyi P, Tudorache I, Gottlieb J, Welte T, Fuehner T. Impact of alpha 1-antitrypsin deficiency and prior augmentation therapy on patients' survival after lung transplantation. Eur Respir J. 2017 Sep 10;50(3):1700962. doi: 10.1183/13993003.00962-2017. Print 2017 Sep. No abstract available. PMID 28890438
- [Result] Cerdan de Las Heras J, Tulppo M, Kiviniemi AM, Hilberg O, Lokke A, Ekholm S, Catalan-Matamoros D, Bendstrup E. Augmented reality glasses as a new tele-rehabilitation tool for home use: patients' perception and expectations. Disabil Rehabil Assist Technol. 2022 May;17(4):480-486. doi: 10.1080/17483107.2020.1800111. Epub 2020 Aug 4. PMID 32750254
- [Result] Patsaki I, Avgeri V, Rigoulia T, Zekis T, Koumantakis GA, Grammatopoulou E. Benefits from Incorporating Virtual Reality in Pulmonary Rehabilitation of COPD Patients: A Systematic Review and Meta-Analysis. Adv Respir Med. 2023 Aug 10;91(4):324-336. doi: 10.3390/arm91040026. PMID 37622840
- [Result] Hayton C, Clark A, Olive S, Browne P, Galey P, Knights E, Staunton L, Jones A, Coombes E, Wilson AM. Barriers to pulmonary rehabilitation: characteristics that predict patient attendance and adherence. Respir Med. 2013 Mar;107(3):401-7. doi: 10.1016/j.rmed.2012.11.016. Epub 2012 Dec 19. PMID 23261311
- [Result] Depew ZS, Novotny PJ, Benzo RP. How many steps are enough to avoid severe physical inactivity in patients with chronic obstructive pulmonary disease? Respirology. 2012 Aug;17(6):1026-7. doi: 10.1111/j.1440-1843.2012.02207.x. PMID 22672739
- [Result] Savci S, Ince DI, Arikan H. A comparison of autogenic drainage and the active cycle of breathing techniques in patients with chronic obstructive pulmonary diseases. J Cardiopulm Rehabil. 2000 Jan-Feb;20(1):37-43. doi: 10.1097/00008483-200001000-00006. PMID 10680096
- [Result] Zisi D, Chryssanthopoulos C, Nanas S, Philippou A. The effectiveness of the active cycle of breathing technique in patients with chronic respiratory diseases: A systematic review. Heart Lung. 2022 May-Jun;53:89-98. doi: 10.1016/j.hrtlng.2022.02.006. Epub 2022 Feb 27. PMID 35235877
- [Result] Barjaktarevic I, Campos M. Management of lung disease in alpha-1 antitrypsin deficiency: what we do and what we do not know. Ther Adv Chronic Dis. 2021 Jul 29;12_suppl:20406223211010172. doi: 10.1177/20406223211010172. eCollection 2021. PMID 34408831
- [Result] Alwadani FA, Wheeler K, Pittaway H, Turner AM. Pulmonary Rehabilitation for Chronic Obstructive Pulmonary Disease Patients with Underlying Alpha-1 Antitrypsin Deficiency: A Systematic Review and Practical Recommendations. Chronic Obstr Pulm Dis. 2024 Jan 25;11(1):121-132. doi: 10.15326/jcopdf.2023.0434. PMID 37813825
- [Result] Nici L, Donner C, Wouters E, Zuwallack R, Ambrosino N, Bourbeau J, Carone M, Celli B, Engelen M, Fahy B, Garvey C, Goldstein R, Gosselink R, Lareau S, MacIntyre N, Maltais F, Morgan M, O'Donnell D, Prefault C, Reardon J, Rochester C, Schols A, Singh S, Troosters T; ATS/ERS Pulmonary Rehabilitation Writing Committee. American Thoracic Society/European Respiratory Society statement on pulmonary rehabilitation. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1390-413. doi: 10.1164/rccm.200508-1211ST. No abstract available. PMID 16760357
- [Result] Crystal RG. Alpha 1-antitrypsin deficiency, emphysema, and liver disease. Genetic basis and strategies for therapy. J Clin Invest. 1990 May;85(5):1343-52. doi: 10.1172/JCI114578. No abstract available. PMID 2185272
- [Result] Nukiwa T, Brantly M, Ogushi F, Fells G, Satoh K, Stier L, Courtney M, Crystal RG. Characterization of the M1(Ala213) type of alpha 1-antitrypsin, a newly recognized, common "normal" alpha 1-antitrypsin haplotype. Biochemistry. 1987 Aug 25;26(17):5259-67. doi: 10.1021/bi00391a008. PMID 2890373
- [Result] Brantly M, Nukiwa T, Crystal RG. Molecular basis of alpha-1-antitrypsin deficiency. Am J Med. 1988 Jun 24;84(6A):13-31. doi: 10.1016/0002-9343(88)90154-4. PMID 3289385
- [Result] DeMeo DL, Silverman EK. Alpha1-antitrypsin deficiency. 2: genetic aspects of alpha(1)-antitrypsin deficiency: phenotypes and genetic modifiers of emphysema risk. Thorax. 2004 Mar;59(3):259-64. doi: 10.1136/thx.2003.006502. PMID 14985567
- [Result] Long GL, Chandra T, Woo SL, Davie EW, Kurachi K. Complete sequence of the cDNA for human alpha 1-antitrypsin and the gene for the S variant. Biochemistry. 1984 Oct 9;23(21):4828-37. doi: 10.1021/bi00316a003. PMID 6093867
- [Result] Lai EC, Kao FT, Law ML, Woo SL. Assignment of the alpha 1-antitrypsin gene and a sequence-related gene to human chromosome 14 by molecular hybridization. Am J Hum Genet. 1983 May;35(3):385-92. PMID 6602546
- [Result] Luisetti M, Seersholm N. Alpha1-antitrypsin deficiency. 1: epidemiology of alpha1-antitrypsin deficiency. Thorax. 2004 Feb;59(2):164-9. doi: 10.1136/thorax.2003.006494. PMID 14760160